CLINICAL TRIAL: NCT01081210
Title: Screening With Pocket-sized Ultrasound of Patients Admitted to Department of Medicine at a Local Hospital
Brief Title: Screening of Patients Admitted to a Local Hospital With Pocket-sized Ultrasound
Status: Completed | Type: Observational
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: LH-2010-1; HD_2009_LU13 (Other: Nord-Trøndelag Health Trust)
Record Dates: First submitted 2010-02-25; First posted 2010-03-05 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Heart Disease; Dyspnea; Aortic Disease; Kidney Disease; Liver Disease
Keywords: Echocardiography; Heart failure; Kidney; Lung; Aorta
MeSH Terms: conditions — Heart Diseases; Dyspnea; Aortic Diseases; Kidney Diseases; Liver Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum blood samples including; hematology, electrolytes, creatinine, liver enzymes and cholestasis parametres, brain natriuretic peptides etc.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ultrasound screening: Patients admitted to Department of medicine at local hospital. Randomized inclusion, informed consent obtained.
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Screening with bedside ultrasound examination
  Other Names: GE Vingmed VScan

SUMMARY:
Ultrasound (US) is widely used as a diagnostic tool in a hospital setting. In a medical department, diagnosis like heart failure or most kinds of heart diseases, hypervolemia, hypovolemia, pleural effusion, pericardial effusion, ascites, diseases in the gall bladder/bile tract, urine tract and venous thrombosis are common. US is the key diagnostic tool in these diagnosis, and on early diagnosis is crucial both on behalf of the patients well-being, and for hospital logistic reasons.

1. The aim is to study the clinical use of pocket sized US as a screening diagnostic tool in an department of internal medicine.

   Method: All patients admitted (in certain preset periods) to Department of medicine will be screened with pocket sized US by expert user. Changes in diagnoses, as well as medications as a result of US screening will be the endpoints. US findings will be validated against standard echocardiography, or standard US/CT/MRI performed at the Radiological department.
2. The aim is to study the clinical use of pocket sized US as a screening diagnostic tool in a department of cardiology.

   Method: All patients admitted (in certain preset periods) to Department of cardiology will be screened with pocket sized US for heart disease, pericardial and pleural effusion. Examinations by expert users. Specific findings could be myocardial dysfunction as heart failure, cardiomyopathies, regional dysfunction due to ischemia, valvular dysfunction, atrial enlargement, and pleural/pericardial effusion. Changes in diagnoses, as well as medications as a result of US screening will be the endpoints. US findings will be validated against standard echocardiography in all.
3. As in 1), but examination by non-expert users compared to expert users.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Dep. of Medicine at Levanger Hospital

Exclusion Criteria:

* Not able to give informed consent

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Dep. of Medicine at Levanger Hospital Randomized study. Both sexes. Age above 16 years
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity | After 3-6 months
  Diagnostic accuracy and clinical usefulness of ultrasound screening as add on examination. Change in working diagnosis after ultrasound examination will be tested, and gold standards (echocardiography and examinations at Department of radiology) will be used for testing of sensitivity and specificity.

SECONDARY OUTCOMES:
Non-experts | After 3-6 months
  Validation of results from ultrasound examination made by non-experts compared to expert users.

CONTACTS AND LOCATIONS:
Overall Officials: Havard Dalen, MD, Principal Investigator — Nord-Trøndelag Health Trust
Locations (2):
- Norway (2):
  - Department of Medicine, Levanger Hospital, Nord-Trøndelag Health Trust, Levanger
  - Levanger Hospital, Department of Medicine, Levanger

REFERENCES:
- [Background] Kimura BJ, Shaw DJ, Agan DL, Amundson SA, Ping AC, DeMaria AN. Value of a cardiovascular limited ultrasound examination using a hand-carried ultrasound device on clinical management in an outpatient medical clinic. Am J Cardiol. 2007 Jul 15;100(2):321-5. doi: 10.1016/j.amjcard.2007.02.104. Epub 2007 May 29. PMID 17631091
- [Background] Roelandt JR. Ultrasound stethoscopy. Eur J Intern Med. 2004 Oct;15(6):337-347. doi: 10.1016/j.ejim.2004.08.002. PMID 15522567
- [Background] Beaulieu Y. Bedside echocardiography in the assessment of the critically ill. Crit Care Med. 2007 May;35(5 Suppl):S235-49. doi: 10.1097/01.CCM.0000260673.66681.AF. PMID 17446784
- [Background] Lucas BP, Candotti C, Margeta B, Evans AT, Mba B, Baru J, Asbury JK, Asmar A, Kumapley R, Patel M, Borkowsky S, Fung S, Charles-Damte M. Diagnostic accuracy of hospitalist-performed hand-carried ultrasound echocardiography after a brief training program. J Hosp Med. 2009 Jul;4(6):340-9. doi: 10.1002/jhm.438. PMID 19670355
- [Background] Martin LD, Howell EE, Ziegelstein RC, Martire C, Whiting-O'Keefe QE, Shapiro EP, Hellmann DB. Hand-carried ultrasound performed by hospitalists: does it improve the cardiac physical examination? Am J Med. 2009 Jan;122(1):35-41. doi: 10.1016/j.amjmed.2008.07.022. PMID 19114170
- [Derived] Andersen GN, Haugen BO, Graven T, Salvesen O, Mjolstad OC, Dalen H. Feasibility and reliability of point-of-care pocket-sized echocardiography. Eur J Echocardiogr. 2011 Sep;12(9):665-70. doi: 10.1093/ejechocard/jer108. Epub 2011 Aug 2. PMID 21810825